CLINICAL TRIAL: NCT06313970
Title: A Multicenter,Open-label,Exploratory Study of QL1706 Plus Nab-paclitaxel and Gemcitabine With or Without Bevacizumab as First-line Treatment in Patients With Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: First-line Regimen With QL1706 Plus Chemo ± Bev in PDAC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-PC-IIT-001
Record Dates: First submitted 2024-03-11; First posted 2024-03-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706+chemotherapy (Experimental): QL1706 administered by intravenous infusion, 5 mg/kg, administered once every 3 weeks, every 3 weeks as a cycle; Albumin paclitaxel administered by intravenous infusion, 125 mg/m2, administered on Days 1 and 8, 1 treatment cycle every 3 weeks; Gemcitabine IV infusion over 30 min, 1000 mg/m2, administered on Days 1 and 8, 1 treatment cycle every 3 weeks; On day 1 of each cycle, drugs were administered in the following order: ql1706 → albumin paclitaxel → gemcitabine.
  The first dose was administered within 2 days of randomization, and subjects used the study drug until protocol-specified criteria for treatment termination were present.
  Interventions: Drug: QL1706; Drug: Nab-paclitaxel; Drug: Gemcitabine
- QL1706+chemotherapy+ bevacizumab (Experimental): QL1706 administered by intravenous infusion, 5 mg/kg, administered once every 3 weeks, every 3 weeks as a cycle; Bevacizumab administered by intravenous infusion, 7.5 mg/kg, administered once every 3 weeks, every 3 weeks as a treatment cycle; Albumin paclitaxel administered by intravenous infusion, 125 mg/m2, administered on Days 1 and 8, 1 treatment cycle every 3 weeks; Gemcitabine IV infusion over 30 min, 1000 mg/m2, administered on Days 1 and 8, 1 treatment cycle every 3 weeks; On day 1 of each cycle, drugs were administered in the following order: ql1706 → bevacizumab → albumin paclitaxel → gemcitabine.
  The first dose was administered within 2 days of randomization, and subjects used the study drug until protocol-specified criteria for treatment termination were present.
  Interventions: Drug: QL1706; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: QL1706 — QL1706 5mg/kg，IV，D1, Q3W
Drug: Nab-paclitaxel — Nab-paclitaxel, 125mg/m2，IV，D1、8, Q3W
Drug: Gemcitabine — gemcitabine，1000mg/m2，IV，D1、8；Q3W.
Drug: Bevacizumab — bevacizumab, 7.5mg/kg，IV，D1；Q3W.
  Arms: QL1706+chemotherapy+ bevacizumab

SUMMARY:
This is a multicenter, open-label, exploratory study to evaluate the efficacy and safety of QL1706 plus nab-paclitaxel and gemcitabine with or without bevacizumab as first-line treatment in patients with unresectable locally advanced or metastatic pancreatic cancer

DETAILED DESCRIPTION:
This study is an open, multicenter, exploratory clinical trial designed to evaluate the efficacy and safety of QL1706 in combination with albumin paclitaxel and gemcitabine with or without bevacizumab for the first-line treatment of patients with unresectable locally advanced or metastatic pancreatic cancer.

The study was conducted in patients with unresectable locally advanced or metastatic pancreatic cancer who had not received prior systemic therapy. Subjects sign informed consent, undergo a screening period of examination and evaluation, which lasts for 21 days, and those who meet the entry criteria enter the treatment period and are randomized 1:1 to receive either QL1706 in combination with albumin paclitaxel and gemcitabine or to receive QL1706 in combination with albumin paclitaxel, gemcitabine, and bevacizumab in 3-week intervals until protocol-specified treatment termination Event. Subjects will be enrolled in the study and will undergo a safety visit prior to D1 dosing for each treatment cycle, please refer to the trial flow chart. Imaging exams and assessments will be performed every 6 weeks (± 7 days) for the first 24 weeks of treatment and every 9 weeks (± 7 days) thereafter until disease progression, initiation of new antitumor therapy, withdrawal of informed consent, or death, whichever occurs first, as confirmed per RECIST v1.1. Additional imaging and evaluation may be performed at any time during the study if clinically indicated.

Subjects will be required to complete safety examinations and imaging assessments at the end of treatment, followed by a safety visit and follow-up until 90 days after the last dose of QL1706 or 30 days after the last dose of other investigational agents, whichever is longer. For subjects who end treatment with non-RECIST v1.1 criteria for disease progression, imaging should be continued to assess time to tumor progression. Survival follow-up is performed after the safety visit, every 60 days (±7 days), to collect and record the subject's survival status and subsequent antitumor therapy.

The study used ORR as the primary endpoint and was planned to enroll 58 subjects, 29 in the QL1706 combined albumin paclitaxel and gemcitabine group and 29 in the QL1706 combined albumin paclitaxel and gemcitabine combined bevacizumab group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study, sign the informed consent form;
2. Age ≥18 years and ≤75 years;
3. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma or adenocarcinoma.
4. Patients have not received prior systemic therapy for unresectable locally advanced or metastatic pancreatic cancer;
5. At least one measurable lesion according to RECIST 1.1 criteria;
6. ECOG Performance Status 0-1;
7. Estimated life expectancy ≥3 months;
8. Adequate major organ function (no medication for blood component, cell growth factor correction therapy is allowed within 14 days before randomization);
9. Women of child-bearing potential must agree to use a reliable, effective method of contraception from the time they provide informed consent until at least 120 days after the last dose of study drug is administered. HCG test must be negative. And must be non-lactating;
10. Male participants whose partner is a woman of child-bearing potential must agree to use a reliable, effective method of contraception from the time they sign an informed consent form until at least 120 days after the last dose of study drug is administered. Male subjects also have to agree not to donate sperm during the same period.

Exclusion Criteria:

1. Histologically or cytologically confirmed other pathological types, such as acinar cell carcinoma, pancreatic neuroendocrine neoplasms or pancreatoblastoma.
2. Patients with other malignant tumors within 5 years, except localized tumor that has been cured;
3. Known active or untreated brain metastases, meningeal metastases, spinal cord compression or leptomeningeal disease.
4. Patients with a history of life-threatening bleeding or a definite risk of bleeding within 6 months before randomization;
5. Has undergone major trauma or surgical treatment within 28 days before randomization or is expected to undergo major surgical treatment during the study period;
6. Poorly controlled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) ；or have a history of hypertensive crisis or hypertensive encephalopathy;
7. Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, pulmonary embolism, etc., occurred within 6 months before randomization;
8. Patients who receive any prior treatments targeting the mechanism of tumor immunity, such as immune checkpoint blockades, immune checkpoint agonists, immune cell therapy, etc.
9. Active autoimmune disease requiring systemic treatment within 2 years before randomization, or autoimmune diseases that may relapse or require scheduled treatment judged by the investigator;
10. Subjects with active hepatitis B or C;
11. Patients with a known history of immunodeficiency or HIV positive;
12. The investigator assessed that it is not appropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 1 years
  ORR is defined as the percentage of subjects with complete response (CR) or partial response (PR) by investigator assessment per RECIST criteria, version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to approximately 1 years
  DCR was defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD).
Duration of Response (DoR) | up to approximately 1 years
  Response will be determined by investigator using RECIST 1.1.
Time to response(TTR) | up to approximately 1 years
  Response will be determined by investigator using RECIST 1.1.
Progression-free survival (PFS) | up to approximately 1 years
  PFS is defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.
Overall survival（OS） | up to approximately 1 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Adverse Events | up to approximately 1 years
  AE assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No